CLINICAL TRIAL: NCT00003281
Title: Phase II Trial of Topotecan and Paclitaxel in Previously Treated Patients With Relapsed Small Cell Lung Cancer
Brief Title: Topotecan and Paclitaxel in Treating Patients With Recurrent or Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-972051; CDR0000066190 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-09-24 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Paclitaxel; Topotecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- topotecan + paclitaxel + radiotherapy (Experimental): Patients receive topotecan IV over 30 minutes on days 1-3 and paclitaxel IV over 3 hours on day 3. Courses repeat every 4 weeks.
  Patients who achieve partial response or stable disease continue treatment in the absence of complete response or disease progression. Patients who develop disease progression in the CNS only should receive whole brain radiotherapy and then continue treatment. Patients who achieve complete remission receive a maximum of 6 courses of treatment. Patients may then undergo prophylactic cranial irradiation and/or thoracic radiotherapy at the discretion at the attending physician.
  Patients are followed every 3 months for 2 years and then at 3 years after study.
  Interventions: Drug: paclitaxel; Drug: topotecan hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: paclitaxel
Drug: topotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of topotecan and paclitaxel in treating patients who have recurrent or refractory small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of combination topotecan and paclitaxel in previously treated patients with small cell lung cancer.
* Determine the response rate and survival in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to length of time since prior treatment (less than 3 months (stratum A) vs 3 months or more (stratum B)). Stratum A closed to accrual effective 06/20/2000.

Patients receive topotecan IV over 30 minutes on days 1-3 and paclitaxel IV over 3 hours on day 3. Courses repeat every 4 weeks.

Patients who achieve partial response or stable disease continue treatment in the absence of complete response or disease progression. Patients who develop disease progression in the CNS only should receive whole brain radiotherapy and then continue treatment. Patients who achieve complete remission receive a maximum of 6 courses of treatment. Patients may then undergo prophylactic cranial irradiation and/or thoracic radiotherapy at the discretion at the attending physician.

Patients are followed every 3 months for 2 years and then at 3 years after study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Stratum A (less than 3 months since prior therapy) closed to accrual effective 06/20/2000)
* Histologically or cytologically confirmed recurrent or refractory small cell lung cancer

  * Only 1 prior regimen allowed (an alternating regimen with cyclophosphamide/doxorubicin/vincristine and etoposide/cisplatin is acceptable)
* No mixed histology
* Measurable or evaluable disease that has not been in the field of prior radiotherapy
* No uncontrolled CNS metastases (treated CNS metastases eligible)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Total bilirubin no greater than 1.5 times upper limit of normal (ULN) OR
* Direct bilirubin normal

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No unstable angina pectoris
* No uncontrolled congestive heart failure
* No myocardial infarction within the past 3 months

Other:

* No uncontrolled infections
* No other concurrent malignancy except skin cancer or localized prostate cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior topoisomerase I inhibitor (e.g., topotecan or irinotecan) or taxane (e.g., paclitaxel or docetaxel)
* At least 3 months since other prior chemotherapy

Radiotherapy:

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* At least 3 weeks since any prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 1998-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 5 years

SECONDARY OUTCOMES:
survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: James R. Jett, MD, Study Chair — Mayo Clinic
Locations (19):
- United States (18):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Dy GK, Jett JR, Geoffroy FJ, Krewer KD, Tazelaar H, Maurer M, Rowland K, Mailliard J, Krook J, Dakhil S, Kutteh L, Kugler J, Wender D. Topotecan and paclitaxel in previously treated patients with relapsed small cell lung cancer: phase II trial of the North Central Cancer Treatment Group. J Thorac Oncol. 2006 Mar;1(3):211-7. doi: 10.1016/s1556-0864(15)31570-7. No abstract available. PMID 17409859